CLINICAL TRIAL: NCT06273566
Title: French Validation of the AdT-Physio Scale for Assessing Adherence and Perception of the Intervention of a Physiotherapist in Patients With Cystic Fibrosis
Brief Title: French Validation of the AdT-Physio Scale
Acronym: Trans-AdT
Status: Recruiting | Type: Observational
Sponsor: Pole Sante Grace de Dieu (Other)
Responsible Party: Sponsor
Other Study IDs: 20230202
Record Dates: First submitted 2024-02-08; First posted 2024-02-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis
Keywords: Translation; Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Participants will have to answer the socio-demographic questions (Age, weight, height, FEV1, FVC) and the AdT-Physio, Brief Cope and GSES questionnaires in random order.

SUMMARY:
The goal of this observational study is to translate and validate the Adt-Physio scale in French, and to validate on a large number of patients the French translation of the Adt-Physio scale as a tool for evaluating adherence and perception of the intervention of a physiotherapist in patients with cystic fibrosis.

participants will have to answer the French trans-AdT scale, the Brief Cope and GSES questionnaire.

DETAILED DESCRIPTION:
Cystic fibrosis is one of the most frequently encountered rare genetic diseases. In 2022, this pathology affected 7,743 people in the French population, i.e. 3% more than in 2021. Previously, this fatal disease only granted a few months of life to child carriers. Today, the median age at death is over 40 years old. The adult population suffering from cystic fibrosis has thus become more numerous than the pediatric population. Among existing treatments, respiratory and musculoskeletal massage physiotherapy occupies a central place in patients' lives. However, the level of adherence to massage physiotherapy is low among young adults (16 to 21 years old) compared to other types of treatments. Faced with epidemiological changes and the daily burden that this chronic pathology represents for those affected, therapeutic adherence should be a major concern for physiotherapists. Indeed, a low level of adherence would increase treatment failures, the risk of premature death, episodes of exacerbations and hospitalizations and would thus reduce quality of life. It is therefore crucial to have means of assessing this parameter in patients with cystic fibrosis. The AdT physio self-assessment questionnaire, validated in Spanish since 2020, has shown clinical validity and reliability for Spanish-speaking patients. Thus, a version of this scale translated and validated in French would offer physiotherapists a relevant tool allowing them to evaluate therapeutic adherence and the perception of their interventions with French-speaking patients suffering from cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

The subjects recruited are patients with cystic fibrosis, over 18 years old, without a lung transplant and able to answer the questionnaires.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects recruited are patients with cystic fibrosis, over 18 years old, without a lung transplant and able to answer the questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
AdT-Physio scale (Adherence to Treatment of Physiotherapy scale) | 1 year
  set of 15 questions divided into two sets, one focusing on patient adherence and the other on beliefs about the treatment and therapist (The total score on the final version of the AdT-Physio scale can range from 14 to 56, in which a high score is indicative of better adherence to physical therapy.)

CONTACTS AND LOCATIONS:
Locations (1):
- PSLA GDD, Caen, France

IPD SHARING:
Plan to Share IPD: No